CLINICAL TRIAL: NCT05201027
Title: A Prospective, Non-comparative, Multicenter Trial to Optimize the IOL Constant of a New Multifocal IOL
Brief Title: Study to Optimize the IOL Constant of a New Multifocal Intraocular Lens
Acronym: HECATE A
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to modify the prototype device used in study
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT ELANA 841P-BER-301-19
Record Dates: First submitted 2022-01-06; First posted 2022-01-21 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Cataract Senile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- trifocal intraocular lens (Experimental): Implantation of new trifocal intraocular lens
  Interventions: Device: trifocal intraocular lens

INTERVENTIONS:
Device: trifocal intraocular lens — cataract extraction and implantation of a posterior chamber trifocal intraocular lens

SUMMARY:
Prospective, non-comparative, multicenter study on medical device with 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient of any gender;
* Patient with clinically significant bilateral age-related cataracts with planned phacoemulsification cataract extraction and suitable for implantation of a posterior chamber trifocal intraocular lens as determined by investigator's medical judgement;
* Projected postoperative corrected distance visual acuity (CDVA) better than 0.2 LogMAR as determined by investigator's medical judgement;
* Preoperative keratometric (corneal) astigmatism ≤1.5 D;
* Clear intraocular media other than cataract;
* Requiring an IOL power within the available range of the investigational IOL (15.0 to +27.0 D, in 0.5 D increments);
* Patient agrees to have surgery of the second eye performed between 1 day and 10 days after the surgery of the first eye.
* Given written informed consent by patient;
* Patient willing and able to comply with examination procedures and schedule for follow-up visits;

Exclusion Criteria:

* Presence of uncontrolled systemic disease that could increase the operative risk or confound the outcome including but not limited to diabetes mellitus, active cancer treatment, mental illness, dementia, immunocompromised, connective tissue disease, clinically significant atopic disease, etc.;
* Ocular condition that may predispose patient to future complications, per investigator's medical judgement, including but not limited to severe dry eye, anterior segment pathology, glaucoma (uncontrolled despite intake of medication), macular degeneration;
* Clinically significant corneal abnormalities, including corneal dystrophy (epithelial, stromal or endothelial dystrophy), irregularity, inflammation or oedema as per Investigator's medical judgement; conditions including but not limited to keratitis, keratoconjunctivitis, kerato uveitis, keratopathy, keratectasia;
* Previous intraocular or corneal/refractive surgery that might confound the outcome of the investigation or increase the risk to the patient (including corneal transplants, removal of pterygium etc.);
* Use of and foreseeable use of systemic medications that may confound the outcome or increase the risk to the patient per investigator's medical judgement (e.g., steroids, Tamsulosin Hydrochloride or other medications including anticholinergics or alpha-adrenergic blocking agents with similar side effects [e.g. small pupil/floppy iris syndrome], anti-metabolites, etc.);
* Patients with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders, optic nerve atrophy etc.) or any other pathologies of the eye that are predicted to cause future acuity loss to 0.2 LogMAR (CDVA) or worse;
* Patients with conditions that increase the risk of zonular rupture during cataract extraction procedure that may affect the postoperative centration or tilt of the lens;
* Patients with previous refractive surgery procedures, including but not limited to LASIK, limbal relaxing incision;
* Planned concomitant ocular procedure during cataract surgery or within the next 6 months (e.g. glaucoma surgery including implantation of MIGS, astigmatic correction surgery, penetrating keratoplasty, laser-assisted in situ keratomileusis);
* Patients who are expected to require retinal laser treatment within the next 6 months per investigator's medical judgement;
* Amblyopia;
* Rubella, congenital, traumatic or complicated cataracts;
* History of or current anterior or posterior segment inflammation, including but not limited to iritis or uveitis;
* Microphthalmos or macrophthalmos;
* Iris defects (e.g. aniridia);
* Optic nerve atrophy;
* Pseudoexfoliation;
* Keratoconus or irregular astigmatism;
* Inability to measure keratometry or biometry (including but not limited to cataract density, patient unable to focus for longer time etc.);
* Pathologic miosis;
* Pregnant, lactating during the course of the investigation, or another condition with associated fluctuation of hormones that could lead to refractive changes;
* Patient whose freedom is impaired by administrative or legal order;
* Concurrent participation in another drug or device investigation that could confound the outcome of this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Optimization of the IOL constant | 6 months
  Optimization of the calculated IOL constant with regression analysis by utilizing the following data measured during the study: Corneal radii, axial length, anterior chamber depth, IOL power, target refraction, manifest refraction and refraction distance

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Quesada, San Salvador, El Salvador